CLINICAL TRIAL: NCT02992028
Title: Randomized Placebo Controlled Trial of Postoperative Pain After Intravenous Vitamin C Injection for Arthroscopic Rotator Cuff Repair
Brief Title: Postoperative Pain After Intravenous Vitamin C Injection for Arthroscopic Rotator Cuff Repair
Acronym: VITCRCR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Himchan Hospital (Other)
Responsible Party: Principal Investigator, Ji Wan Park, Director, Himchan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HCH 112294-01-201610-01
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff repair; Vitamin C; postoperative pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative | interventions — Vitamins; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous vitamin C injection (Experimental): During the first 30 min after beginning of the rotator cuff repair, treatment group received infusion of 3 g vitamin C (ascorbic acid) in 500 ml of Ringer.
  Interventions: Drug: Intravenous Nutrition (Vitamins) injection
- Intravenous saline injection (Placebo Comparator): During the first 30 min after beginning of the rotator cuff repair, sham group received 6 ml normal saline in 500 ml of Ringer.
  Interventions: Drug: Intravenous Saline injection

INTERVENTIONS:
Drug: Intravenous Nutrition (Vitamins) injection
  Other Names: Preoperative Vitamin C injection
  Arms: Intravenous vitamin C injection
Drug: Intravenous Saline injection
  Other Names: Preoperative Saline injection
  Arms: Intravenous saline injection

SUMMARY:
1. Treatment of rotator cuff tear The rotator cuff tear is the most demanding part of the shoulder surgery. Rotator cuff degeneration is thought to be the largest cause of rotator cuff tear.

   As the field of shoulder surgery evolves, the diagnosis and surgical treatment of the rotator cuff tear was increased. Repair and reconstruction of the rotator cuff tear annually more than 300,000 have been performed according to US statistics.

   Rotator cuff repair is a successful procedure, both objectively and subjectively, with regard to pain relief and functional outcome.
2. postoperative pain management after rotator cuff repair Shoulder surgeries are associated with a level of postoperative pain requiring opioid use for several days. The opioid requirements after shoulder surgery have been reported to be similar to those required after gastrectomy or thoracotomy, which might cause several opioid-related side effects, such as nausea and vomiting, pruritus, urinary distention, and constipation. Although the introduction of arthroscopy has reduced postoperative pain, a considerable proportion of patients suffer from moderate to severe acute postoperative pain, as its benefit is typically apparent after a few days. Consequently, proactive pain control is also required during the first 24-48 h after arthroscopic shoulder surgeries, just like in open surgeries. Adequate pain management during the immediate postoperative period is not only important for patient satisfaction and well-being, but also for facilitating postoperative rehabilitation and preventing persistent postsurgical pain.

Recently preoperative intravenous vitamin C has shown to increase the analgesic effect after otorhinolaryngologic surgery and thoracic surgery. Vitamin C is a water-soluble and known to have anti oxidant action, and fewer side effects.

However, there is no report about the analgesic effect of vitamin C after arthroscopic rotator cuff repair.

The purpose of this trial was to compare the effects of a intravenous vitamin C injection on postoperative pain and opioid consumption versus non-treated group after arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff tear patients undergoing arthroscopic rotator cuff tear

Exclusion Criteria:

* age <45 or >80
* allergies to medications used in the study
* history of renal diseases, a coagulation abnormality, a hepatic disease, or drug abuse
* definite radiographic evidence of osteoarthritis of the glenohumeral joint
* inflammatory arthritis including rheumatoid arthritis
* a history of acute trauma
* systemic conditions associated with chronic pain
* a history of infection
* an inability to understand the questionnaires

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Recorded at 24 hours after surgery
  from 0mm to 100mm in 10-mm increments (indicating no pain or extreme pain)

SECONDARY OUTCOMES:
Postoperative narcotic consumption | up to postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ji Wan Park, M.D., Study Chair — Himchan Hospital
Locations (1):
- Himchan Hopital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Sadeghpour A, Alizadehasl A, Kyavar M, Sadeghi T, Moludi J, Gholizadeh F, Totonchi Z, Ghadrdoost B. Impact of vitamin C supplementation on post-cardiac surgery ICU and hospital length of stay. Anesth Pain Med. 2015 Feb 19;5(1):e25337. doi: 10.5812/aapm.25337. eCollection 2015 Feb. PMID 25789244
- [Background] Jo CH, Shin JS, Huh J. Multimodal analgesia for arthroscopic rotator cuff repair: a randomized, placebo-controlled, double-blind trial. Eur J Orthop Surg Traumatol. 2014 Apr;24(3):315-22. doi: 10.1007/s00590-013-1208-z. Epub 2013 Mar 14. PMID 23494779
- [Background] Jeon Y, Park JS, Moon S, Yeo J. Effect of Intravenous High Dose Vitamin C on Postoperative Pain and Morphine Use after Laparoscopic Colectomy: A Randomized Controlled Trial. Pain Res Manag. 2016;2016:9147279. doi: 10.1155/2016/9147279. Epub 2016 Oct 30. PMID 27872555
- [Background] Ayatollahi V, Dehghanpour Farashah S, Behdad S, Vaziribozorg S, Rabbani Anari M. Effect of intravenous vitamin C on postoperative pain in uvulopalatopharyngoplasty with tonsillectomy. Clin Otolaryngol. 2017 Feb;42(1):139-143. doi: 10.1111/coa.12684. Epub 2016 Jun 7. PMID 27219124
- [Background] Hasanzadeh Kiabi F, Soleimani A, Habibi MR, Emami Zeydi A. Can vitamin C be used as an adjuvant for managing postoperative pain? A short literature review. Korean J Pain. 2013 Apr;26(2):209-10. doi: 10.3344/kjp.2013.26.2.209. Epub 2013 Apr 3. No abstract available. PMID 23614091
- [Background] Coghlan JA, Forbes A, Bell SN, Buchbinder R. Efficacy and safety of a subacromial continuous ropivacaine infusion for post-operative pain management following arthroscopic rotator cuff surgery: a protocol for a randomised double-blind placebo-controlled trial. BMC Musculoskelet Disord. 2008 Apr 22;9:56. doi: 10.1186/1471-2474-9-56. PMID 18430210